CLINICAL TRIAL: NCT00344461
Title: Cell Cycle Independent Antiretroviral Therapy: Combination of Nevirapine, FTC, and Tenofovir
Brief Title: A Two Year Study of the Clinical Efficacy of the Combination of Emtricitabine, Tenofovir, and Nevirapine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-23783
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV
MeSH Terms: interventions — Nevirapine; Racivir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nevirapine, FTC, Tenofovir (Experimental): Open Label Drugs- Nevirapine 200 mg twice a day, FTC 200 mg once a day and Tenofovir 300 mg once a day for 96 weeks.
  Interventions: Drug: Nevirapine, FTC, and Tenofovir

INTERVENTIONS:
Drug: Nevirapine, FTC, and Tenofovir — One arm only - Open label using FTC 200 mg p.o. qd, and Tenofovir 300 mg p.o. qd, and Nevirapine 200 mg b.i.d.

SUMMARY:
Open label, two year study of the clinical efficacy of the combination of FTC, Tenofovir, and Nevirapine. Sixty HIV infected patients without previous exposure to antiretroviral therapy will be enrolled. Study will include a pharmacokinetic substudy to evaluate the interaction of FTC and Nevirapine. Truvada may be used.

DETAILED DESCRIPTION:
Description of study design This is an open-labeled clinical trial evaluating an antiretroviral treatment regimen in which the drugs have demonstrated in vitro activity in both, resting and activated mononuclear cells. These drugs include: FTC 200 mg p.o. qd, and Tenofovir 300 mg p.o. qd, and Nevirapine 200 mg b.i.d.

Eligible patients must be at least 18 years of age, be referred by their primary HIV provider for antiretroviral therapy or if the patient is self referred, have a cluster of differentiation 4 (CD4) cell count of < 250/mm3 and have a viral load >5,000c/ml. Eligibility requirement for women is that they must have a CD4 cell count of <250 at the time of enrollment. This cutoff for women is based on unpublished data that there may be increased hepatotoxicity in women with a CD4 cell count > 250 cell/mm3. The screening evaluation will take place the day the informed consent is signed. During that screening evaluation, the patient will undergo a history and physical examination, and will have study labs drawn. Within 60 days of the screening evaluation and meeting all eligible criteria, the patient will be placed on the study treatment regimen. Patients will be evaluated at the clinic on Day 0 (therapy initiation), weeks 2, 4, 6, 8, 12, 16, and then every 8 weeks until 48 weeks and thereafter every 12 weeks through week 96. At the end of the study, all patients may continue their current antiretroviral treatment regimen at the discretion of the patient and their primary care provider.

Pharmacokinetic Analysis Sub Study A pharmacokinetic evaluation will be performed in first 7 volunteers to assess the impact of FTC on Nevirapine and vice versa. Pharmacokinetic analysis will be performed at end of week 2 ( day 14) during 200mg qd start up period. Samples will be obtained at baseline and 1, 3, 6, 12 and 24 hours post Nevirapine dosing. Pharmacokinetic analysis will be repeated at the week 8 visit. Samples will be obtained at baseline and 1, 3, 6, 12 and 24 hours post Nevirapine.

Assignment of patients There will be 60 patients involved in this clinical trial. This is an open-labeled study. There are no placebos involved in this study.

Dose and dose selection The dosages of medications are those that are currently used as standard clinical practice: Nevirapine 200 mg b.i.d. (1-200 mg tablet b.i.d.); Emtricitabine (FTC) 200mg po qd.(1-200mg capsule); Tenofovir 300 mg once-a-day (1-300 mg tablet qd).

Justification of study design All study patients require treatment for their HIV infection. All of the drugs used in this study are FDA-Approved. Tenofovir and FTC are approved as a once-a-day treatment medication. Nevirapine (NVP) is approved for BID dosing.

NOTE: That whenever Nevirapine is being prescribed, there will be a lead-in period of 14 days in which Nevirapine will be prescribed as 200 mg once a day followed by 200 mg BID as is the recommended standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit, and confirmed by Western blot, positive HIV-1 blood culture, positive HIV serum antigen, or plasma viremia at any time prior to study entry. If no record exists, testing must occur at screening.
2. Male or female, age 18 to 75 years of age.
3. Able to sign the informed consent, and is willing to comply with the requirements of this clinical trial.
4. Available for at least 96 weeks of follow up.
5. Males: deemed a candidate for antiretroviral therapy per referring primary care provider. (If patient is self referred, CD4 cell count must be <400 cells/mm3 and viral load>5,000c/ml) Females: CD4 cell count must be less than 250 cells/mm3 and viral load >5,000 c/mL at time of enrollment.
6. If female and of child bearing potential must consent to using at least two forms of contraception.
7. Participants will be "treatment naive" as no prior antiretroviral therapy or antiretroviral therapy for less than 7 days in the past.

Exclusion Criteria:

1. Evidence of mutation associated with primary drug resistance to Nevirapine (K103N, Y181C, Y188L, G190S), Tenofovir (M41L, T69 insertion, Q151M, L210W,and K65R), and/or FTC (184V) previously documented, or at time of screening.
2. Patients with any of the following laboratory parameters at the screening visit: estimated creatinine clearance of <60 ml/min; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times the upper limits of normal; total bilirubin >1.5 mg/dL.
3. Women with CD4 cell count > 250 cells/ mm3 at time of entry or in males with a CD4 cell count less than 400/mm3, along with a viral load greater than 5,000c/ml. for both males and females.
4. Pregnant women or women who are breast feeding.
5. Unwillingness to use effective barrier contraception.
6. Patients with current alcohol abuse or illicit drug use that in the opinion of the Principal Investigator may interfere with the patient's ability to comply with the protocol requirements.
7. Patients with malabsorption or severe chronic diarrhea for more than 30 days.
8. Current treatment for malignancy other than basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
9. History of any chronic illness or other condition that in the opinion of the investigator would interfere with the conduct or completion of the study.
10. Patient who is, in the opinion of the investigator, unable to complete the 96-week dosing period and protocol evaluations and assessments.
11. Experimental vaccines, to include HIV vaccines.
12. Patient who is currently enrolled in an experimental protocol, or is receiving an experimental medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Redfield, MD, Principal Investigator — University of Maryland, School of Medicine, IHV; Charles E Davis, MD, Principal Investigator — University of Maryland, School of Medicine, IHV
Locations (1):
- University of Maryland, Institute of Human Virology, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Amoroso A, Gilliam BL, Talwani R, Boyce C, Redfield RR, Davis CE. Viral load decay in antiretroviral-naive patients receiving once-daily tenofovir and emtricitabine plus twice-daily nevirapine. HIV Clin Trials. 2009 Sep-Oct;10(5):320-3. doi: 10.1310/hct1005-320. PMID 19906624

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Group (TDF/FTC & NVP): To evaluate the long-term antiviral activity of a three cell cycle independent reverse transcriptase regimen consisting of Nevirapine 200mg twice-a-day, Tenofovir 300mg and Emtricitabine 200mg once-a-day in the treatment of patients with chronic HIV infection.
Period: Overall Study
Arm/Group | Single Group (TDF/FTC & NVP)
Started | 54
Completed | 33
Not Completed | 21
Not completed — Adverse Event | 6
Not completed — Death | 1
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- TDF, FTC & NVP: To evaluate the long-term antiviral activity of a three cell cycle independent reverse transcriptase regimen consisting of Nevirapine 200mg twice-a-day, Tenofovir 300mg and Emtricitabine 200mg once-a-day in the treatment of patients with chronic HIV infection.
Arm/Group | TDF, FTC & NVP
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 51
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response
Description: The primary outcome is sustained Virologic response, defined as HIV-1 RNA <500 copies/mL until trial completion at 96 weeks.
Time Frame: 96 Weeks
Population: HIV-1 infected Males: cluster of differentiation 4 (CD4) cell count less than 400 cells/mm3 and viral load greater than 5,000c/ml) Females: CD4 cell count less than 250 cells/mm3 and viral load greater than 5,000 c/mL at time of enrollment. Treatment naive
Measure: Count of Participants; unit: Participants
Arm/Group | Single Group (TDF/FTC & NVP)
Number analyzed (Participants) | 54
Participants | 33

2. Secondary Outcome: Patients With Grade 2, 3 and 4 Adverse Events and Laboratory Toxicities
Description: The number of participants with grades 2,3 and 4 adverse events and laboratory toxicities.
Time Frame: Protocol length is 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nevirapine, FTC, Tenofovir
Number analyzed (Participants) | 54
Participants | 13

3. Secondary Outcome: Patients With Plasma HIV RNA < 50 Copies/mL
Description: The number of participants with plasma HIV RNA < 50 copies/mL
Time Frame: 96 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Group (TDF/FTC & NVP)
Number analyzed (Participants) | 54
Participants | 32

4. Secondary Outcome: Patients With Plasma HIV RNA < 400 Copies/mL
Description: The number of participants with plasma HIV RNA < 400 copies/mL
Time Frame: 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nevirapine, FTC, Tenofovir
Number analyzed (Participants) | 54
Participants | 32

5. Secondary Outcome: Change in Plasma HIV RNA From Baseline to Week 96
Description: Percent Change From Baseline in Plasma HIV RNA at 96 weeks
Time Frame: Baseline to week 96
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Nevirapine, FTC, Tenofovir
Number analyzed (Participants) | 54
percentage of change | 3.32 (.043)

6. Secondary Outcome: Changes in CD4 Cell Count From Baseline and Week 96
Description: To determine the mean change from Baseline in CD4 cell count to week 96.
Time Frame: Baseline to week 96
Measure: Mean (Standard Deviation); unit: percentage of CD4 Increase
Arm/Group | Nevirapine, FTC, Tenofovir
Number analyzed (Participants) | 54
percentage of CD4 Increase | 252 (89.91)

ADVERSE EVENTS:
Time Frame: 96 weeks
Description: A written report will be filed with the Institutional Review Board (IRB) within 5 working days for serious adverse event and annually for all others.
Groups:
- FTC, TDF, & NVP: To evaluate the long-term antiviral activity of a three cell cycle independent reverse transcriptase regimen consisting of Nevirapine 200mg twice-a-day, Tenofovir 300mg and Emtricitabine 200mg once-a-day in the treatment of patients with chronic HIV infection.
Arm/Group | FTC, TDF, & NVP
All-Cause Mortality (participants affected / at risk) | 1/54
Serious Adverse Events (participants affected / at risk) | 16/54
Other Adverse Events (participants affected / at risk) | 13/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FTC, TDF, & NVP (N=54)
Neutrapenia (Blood and lymphatic system disorders) | 2 (2)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
Grade 3 & 4 Liver Function Test (Hepatobiliary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Grade 4 alanine aminotransferase (ALT) test (Hepatobiliary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Stevens Johnson
CMV Retinitis (Eye disorders) | 1 (1)
Malignant Lymphoma (Blood and lymphatic system disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1)
Diffused Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right Femoral Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FTC, TDF, & NVP (N=54)
Syncopy (General disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Sinusitis (General disorders) | 1 (1)
Drug Detoxicity (General disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Herpes Zoster Othalmicus (Eye disorders) | 1 (1)
Left Hand Trauma (General disorders) | 1 (1)
Stabbing (General disorders) | 1 (1)
Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Preseptal Cellulitis (Eye disorders) | 1 (1)
Viral Syndrome (Infections and infestations) | 1 (1)
Abscess Right Leg (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No